CLINICAL TRIAL: NCT04128891
Title: PRospectIve Study of Sacubitril/ValsarTan on MyocardIal OxygenatioN and Fibrosis in PatiEnts With Heart Failure and Preserved Ejection Fraction
Brief Title: Study of Sacubitril/ValsarTan on MyocardIal OxygenatioN and Fibrosis in Heart Failure With Preserved Ejection Fraction
Acronym: PRISTINE-HF
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding not approved
Sponsor: Flinders University (Other)
Responsible Party: Principal Investigator, Joseph Selvanayagam, Professor, Flinders University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FlindersU
Record Dates: First submitted 2019-08-21; First posted 2019-10-16 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacubitril/Valsartan (Experimental): 30 participants to be administered Sacubitril/Valsartan (Entresto) tablets, minimum dose of 49/51mg or maximum dose of 97/103 mg twice daily for the duration of the study (two years).
  Interventions: Drug: Sacubitril-Valsartan
- Valsartan (Active Comparator): 30 participants to be administered Valsartan tablets, minimum dose 80 mg or maximum dose of 160 mg twice daily for the duration of the study (two years).
  Interventions: Drug: Sacubitril-Valsartan

INTERVENTIONS:
Drug: Sacubitril-Valsartan — Cardiomagnetic Resonance Imaging
  Other Names: Valsartan

SUMMARY:
To assess the effect of ARNI on myocardial deoxygenation at stress and myocardial fibrosis, and correlate this to changes in myocardial systolic and diastolic function in HFpEF patients.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is increasing in incidence and accounts for one third to one half of all heart failure admissions worldwide. It portrays a significant burden in terms of prevalence, morbidity and mortality. It is a complex clinical syndrome characterized by multiple pathophysiological mechanisms affecting the cardiac structure and function culminating to increased ventricular filling pressures. The definition of HFpEF remains an evolving concept and the exact definition by various learned societies is not uniform. The recent ANZ heart failure guidelines defines HFpEF as the presence of typical symptoms with or without signs of heart failure, with a measured left ventricular ejection fraction of at least 50% and objective evidence of relevant structural heart disease or diastolic dysfunction without an alternative cause. Despite some common clinical features, there is heterogeneity in the causes of HFpEF, and it is likely that it represents a broad cohort of patients with a range of comorbid conditions. In addition to clinical variability, there is morphological and functional variability at the myocardial level. For instance, whilst left ventricular hypertrophy and left atrial dilatation are traditionally considered morphological hallmarks, they are not universally present, and one third to one half of patients do not demonstrate one or both of these features. Furthermore whilst diastolic dysfunction is considered a sine qua non of the disease, and is recognised in the current guidelines, up-to one third of HFpEF patients in echocardiographic sub-studies have normal diastolic function even in the presence of elevated natriuretic peptides.

The heterogeneous phenotypes in HFpEF have potentially confounded previous trials. Therefore, the identification of various structural phenotypes capable of segmenting the HFpEF population into relevant pathophysiologic categories represents a promising approach. Post-mortem endomyocardial biopsy studies from HFpEF patients have suggested that some of the cardiac structural phenotypes are related to myocyte hypertrophy, interstitial fibrosis, myocardial inflammation due to oxidative stress and epicardial coronary artery disease. In addition, a better understanding of the mechanisms that contribute to the pathophysiology of HFpEF is emerging from pre-clinical, interventional and mechanistic studies. In HFpEF, proinflammatory cardiovascular and non-cardiovascular coexisting conditions (e.g., hypertension, obesity) lead to systemic microvascular endothelial inflammation. This results in myocardial inflammation and fibrosis, increases in oxidative stress and alterations in cardiomyocyte signalling pathways. These alterations promote cardiomyocyte remodeling and dysfunction as well as coronary microvascular dysfunction. A recent study showed that there is a high prevalence of coronary microvascular dysfunction in HFpEF even in the absence of unrevascularized macrovascular coronary artery disease and was correlated with markers of heart failure severity.

Cardiac imaging is pivotal in the evaluation of patients with suspected HFpEF. 2D Echocardiography is able to non-invasively measure left ventricular systolic and diastolic dysfunction, as well as characterise left ventricular filling pressures. Echocardiographic data adds incremental prognostic information in patients with HFpEF. These include assessment of left ventricular hypertrophy, left atrial volume, E/e' ratio, tricuspid regurgitation velocity, right ventricular function and global longitudinal strain. However, echocardiography is unable to easily characterise myocardial tissue nor assess myocardial microvascular function. The application of Cardiovascular Magnetic Resonance (CMR) imaging is increasingly recognised and is currently the standard modality for assessing atrial / ventricular volumes, quantifying ejection fraction and left ventricular mass. It is uniquely able to provide information on morphology, function, perfusion, viability, and tissue characterization in a single examination. Hence, CMR is an ideal tool to delineate the various cardiac structural phenotypes that have been described in HFpEF patients. In addition to routinely used CMR parameters, there are a number of emerging CMR applications that have the potential in advancing our understanding of HFpEF. The important amongst them are the assessment of myocardial oxygenation using Oxygen Sensitive CMR (OS-CMR) and diffuse myocardial fibrosis using T1 mapping. OS-CMR can directly assess the myocardial tissue oxygenation and potentially measure mismatches in myocardial oxygen demand and supply. OS-CMR is based on the principle of changes of paramagnetic properties of haemoglobin due to the effects of oxygenation. The change from oxygenated to de-oxygenated haemoglobin leads to a change in the magnetic resonance signal intensity (SI). An increased myocardial de-oxygenation is reflected as a drop in SI on the T2 weighted CMR images. Hence, this allows in vivo assessment of myocardial ischaemia at the tissue level, relying on accumulation of de-oxyhaemoglobin following vasodilator stress. The change in SI is quantified as a percentage of signal change. Myocardial fibrosis has been implicated in the pathophysiology of HFpEF. Both focal replacement fibrosis and interstitial fibrosis promote adverse ventricular remodelling in HFpEF. The pattern of interstitial fibrosis is diffuse in HFpEF and cannot be detected using the late gadolinium enhancement technique. Recent improvements in parametric mapping techniques (such as T1, T2 and T2*) has made non-invasive assessment of diffuse interstitial and fibrotic changes clinically feasible. CMR T1 parametric mapping techniques enable quantification of the extracellular volume (ECV), a surrogate marker of diffuse fibrosis, and have been validated histologically. Hence it is possible that CMR along with OS-CMR, parametric imaging and late gadolinium enhancement represents the ideal non-invasive modality to study and understand the various pathophysiological mechanisms in HFpEF patients.

A number of biomarkers associated with heart failure are well recognized and measuring their concentrations in circulation can provide valuable information about the diagnosis, prognosis, and management. These biomarkers have significantly enhanced the understanding of the pathophysiology of HFpEF, however only a few are currently being used in clinical practice. The measurement of natriuretic peptides (BNP or NT-proBNP) is recommended by current guidelines as they provide incremental value. Cardiac troponin testing is recommended to establish prognosis in acute heart failure and may be used for prognostication in chronic heart failure as well. Novel biomarkers are increasingly becoming validated and recognized in the care of patients with heart failure. These include galectin-3, ST2, renin and cGMP and they alter in response to cardiac remodelling and fibrosis. However, the role of these biomarkers in microvascular dysfunction has not been systematically studied in HFpEF.

Currently, there are no proven pharmacological therapies for patients with HFpEF. This is evident on HFpEF patients trial on beta-blockers, calcium channel blockers, angiotensin converting enzyme inhibitors, and angiotensin receptor blockers which have failed to demonstrate a significant clinical benefit. The first-in-class angiotensin receptor neprilysin inhibitor (ARNI) sacubitril/valsartan holds promise based on its pharmacodynamic profile. It simultaneously blocks the renin-angiotensin-aldosterone system and the endopeptidase neprilysin. Neprilysin is a ubiquitous enzyme that is responsible for the breakdown of many vasoactive peptides, including the biologically active natriuretic peptides. Sacubitril/valsartan has reduced cardiovascular and all-cause mortality in patients with heart failure and reduced ejection fraction, compared with enalapril. In addition, the biomarkers associated with profibrotic signalling are significantly decreased with ARNI therapy in patients with reduced ejection fraction. In HFpEF patients, the PARAMOUNT-HF Phase II trial has demonstrated significant reduction of NT-proBNP with ARNI in comparison with Valsartan.However, in the recently published PARAGON-HF trial, sacubitril/valsartan did not result in a significantly lower rate of total hospitalizations for heart failure and death from cardiovascular causes among patients with HFpEF. In patients with HFpEF, the effect of ARNI therapy on the various emerging pathophysiological mechanisms remains unknown. Myocardial fibrosis is an important pathophysiological mechanism in HFpEF. Treatment options to block or reverse fibrosis in HFpEF have proven elusive. Angiotensin-receptor blockers have been shown to induce regression of severe myocardial fibrosis in hypertensive patients. In mouse models, ARNI ameliorates maladaptive cardiac remodeling and fibrosis in pressure overload-induced hypertrophy. Although not approved for use in HFpEF, ARNI is an attractive option to mitigate myocardial hypertrophy, fibrosis, ischaemia, and impaired ventricular-arterial coupling, which are all closely related to increased left ventricular filling pressures, a common hallmark of this multifaceted syndrome.

Thus, there remains an enormous unmet need for effective therapy in the group of HFpEF patients. HFpEF is a heterogeneous syndrome, with different degrees of contribution from various pathophysiological processes. In patients with HFpEF, the effect of ARNI therapy on the various postulated structural phenotypes remain unexplored. ARNI has the potential to reduce both ischaemia and fibrosis, and both can be accurately measured utilizing CMR. Therefore, by combining CMR with echocardiography, the investigators aim to assess the effect of ARNI on myocardial deoxygenation at stress and myocardial fibrosis, and correlate this to changes in myocardial systolic and diastolic function in HFpEF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent will be obtained before any assessment is performed
2. ≥ 40 years of age, male or female
3. LVEF ≥45% by echocardiography during the screening period
4. Symptom(s) of heart failure requiring treatment with diuretic(s) for at least 30 days prior to screening visit
5. Current symptom(s) of heart failure (NYHA functional class II to IV)
6. Structural heart disease evidenced by at least 1 of the following echocardiography findings:

   1. Left atrial (LA) enlargement defined by at least 1 of the following: LA width (diameter) ≥3.8 cm or LA length ≥5.0 cm or LA area ≥20 cm2 or LA volume ≥55 ml or LA volume index ≥29 ml/m2
   2. Left ventricular hypertrophy defined by septal thickness or posterior wall thickness ≥1.2 cm
7. Elevated NT-proBNP (atleast 1 of the following)

   1. NT-proBNP >300 pg/ml for patients not in atrial fibrillation or >900 pg/ml for patients in atrial fibrillation during initial screening
   2. Heart failure hospitalization (defined as heart failure listed as the major reason for hospitalization) within 9 months prior to screening visit and NT-proBNP >200 pg/ml for patients not in atrial fibrillation or >600 pg/ml for patients in atrial fibrillation during initial screening

Exclusion Criteria:

1. Any prior echocardiographic measurement of LVEF <45%
2. Acute coronary syndrome (including myocardial infarction), cardiac surgery, other major cardiovascular surgery, or percutaneous coronary intervention within 3 months
3. Known unrevascularized epicardial coronary artery disease (> 50% stenosis in any major epicardial coronary artery)
4. Current acute decompensated heart failure requiring augmented therapy with intravenous diuretic agents, vasodilator agents, and/or inotropic drugs
5. Patients who require treatment with 2 or more of the following: an angiotensin converting enzyme inhibitor, an angiotensin receptor blocker, or a renin inhibitor
6. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
7. Patients with a known history of angioedema
8. Probable alternative diagnoses that in the opinion of the investigator could account for the patient's heart failure symptoms such as significant pulmonary disease (including primary pulmonary hypertension), anaemia, or obesity. Specifically, patients with the following are excluded:

   1. Severe pulmonary disease including chronic obstructive pulmonary disease (i.e., requiring home oxygen therapy, chronic oral steroid therapy or hospitalized for pulmonary decompensation within 12 months) or
   2. Haemoglobin <10 g/dl, or
   3. Body mass index >40 kg/m2
9. Patients with any of the following:

   1. Systolic blood pressure (SBP) ≥180 mm Hg at entry, or
   2. SBP >150 mm Hg and <180 mm Hg at entry unless the patient is receiving 3 or more antihypertensive drugs.
   3. SBP <110 mm Hg at entry
10. Current participation in another investigational drug or device.
11. Patients with history of any dilated cardiomyopathy, including peripartum cardiomyopathy, chemotherapy-induced cardiomyopathy, or viral myocarditis
12. Evidence of right-sided heart failure in the absence of left-sided structural heart disease
13. Known pericardial constriction, genetic hypertrophic cardiomyopathy, or infiltrative cardiomyopathy
14. Clinically significant congenital heart disease that could be the cause of the patient's symptoms and signs of heart failure
15. Presence of hemodynamically significant valvular heart disease in the opinion of the investigator
16. Stroke, transient ischemic attack, carotid surgery, or carotid angioplasty within the 3 months
17. Carotid artery disease or valvular heart disease likely to require surgical or percutaneous intervention during the trial
18. Life-threatening or uncontrolled dysrhythmia, including symptomatic or sustained ventricular tachycardia and atrial fibrillation or atrial flutter with a resting ventricular rate >110 beats per minute
19. Patients with a cardiac resynchronization therapy device
20. Patients with prior major organ transplant or intent to transplant (i.e., on transplant list)
21. Any surgical or medical condition that in the opinion of the investigator may place the patient at higher risk from his/her participation in the study or is likely to prevent the patient from complying with the requirements of the study or completing the study
22. Any surgical or medical condition that might significantly alter the absorption, distribution, metabolism, or excretion of study drugs, including but not limited to any of the following: any history of pancreatic injury, pancreatitis, or evidence of impaired pancreatic function/injury within the past 5 years
23. Evidence of hepatic disease as determined by any 1 of the following: SGOT (AST) or SGPT (ALT) values exceeding 3× the upper limit of normal, bilirubin >1.5 mg/dl at entry
24. Patients with severe renal impairment of the following: eGFR <30 ml/min/1.73 m2 as calculated by the Modification in Diet in Renal Disease (MDRD) formula at entry
25. Presence of known functionally significant bilateral renal artery stenosis
26. Patients with serum potassium >5.2 mmol/l (mEq/l) at entry
27. History or presence of any other disease with a life expectancy of <3 years
28. History of noncompliance to medical regimens and patients who are considered potentially unreliable
29. History or evidence of drug or alcohol abuse within the past 12 months
30. Persons directly involved in the execution of this protocol
31. History of malignancy of any organ system (other than localized basal or squamous cell carcinoma of the skin or localized prostate cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
32. Pregnant or nursing (lactating) women
33. Women of child-bearing potential
34. Contraindications to CMR (claustrophobia, implanted medical devices like pacemakers / defibrillators, cochlear implants, intracranial clips, iron fragments in eyes, inability to lie flat for the scanning period)
35. Contraindications to Gadolinium (eGFR <30 ml/min/1.73 m2 as calculated by the MDRD formula at entry or previous know serious allergy)
36. Contraindications to Adenosine (second or third-degree atrioventricular block, asthma, concurrent dipyridamole use)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
• To study the effects of Sacubitril/Valsartan on microvascular function and ischaemia in HFpEF patients. | 12 Months
  The HFpEF participants on Sacubitril/valsartan with improvement in microvascular function and ischaemia, as assessed by OS-CMR at rest and stress (ΔSI: signal intensity change, at baseline and at 12 months).

SECONDARY OUTCOMES:
2.1 Incidence of microvascular dysfunction in HFpEF | 12 Months
  The proportion of HFpEF patients with microvascular dysfunction, as assessed by OS-CMR ΔSI.
2.2 Extent of myocardial fibrosis in HFpEF | 12 Months
  Baseline assessment of myocardial fibrosis in HFpEF patients and assess the response to Sacubitril/Valsartan by measuring changes in myocardial ECV
2.3 Assessment of left ventricular diastolic function in HFpEF | 12 Months
  Baseline echocardiographic assessment of left ventricular diastolic function in HFpEF patients and assess the response to Sacubitril/Valsartan.
2.4 New York Heart Association (NYHA) class | 12 Months
  Baseline evaluation of NYHA class and change in NYHA class at 12 months following Sacubitril/Valsartan therapy.
2.5 Functional assessment | 12 Months
  Baseline computation of functional status by 6-minute walk test and evaluate the response to Sacubitril/Valsartan therapy
2.6 Number of heart failure related hospitalisations | 12 Months
  The number of HFpEF patients admitted with heart failure during the study period.
2.7 Cardiac mortality | 12 Months
  Cardiac mortality during the study period
2.8 All-cause mortality. | 12 Months
  All-cause mortality during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Carmine De Pasquale, Assoc Prof, Principal Investigator — Flinders Medical Centre; Majo Joseph, Doctor, Principal Investigator — Flinders Medical Centre; Rajiv Ananthakrishna, Doctor, Principal Investigator — Flinders Medical Centre; Michael Stokes, Doctor, Principal Investigator — Royal Adelaide Hospital; Sean Lal, Doctor, Principal Investigator — Royal Prince Alfred; David Kaye, Professor, Principal Investigator — Baker Institute/ Alfred Hospital

REFERENCES:
- [Background] Fonarow GC, Stough WG, Abraham WT, Albert NM, Gheorghiade M, Greenberg BH, O'Connor CM, Sun JL, Yancy CW, Young JB; OPTIMIZE-HF Investigators and Hospitals. Characteristics, treatments, and outcomes of patients with preserved systolic function hospitalized for heart failure: a report from the OPTIMIZE-HF Registry. J Am Coll Cardiol. 2007 Aug 21;50(8):768-77. doi: 10.1016/j.jacc.2007.04.064. Epub 2007 Aug 6. PMID 17707182
- [Background] Lam CS, Donal E, Kraigher-Krainer E, Vasan RS. Epidemiology and clinical course of heart failure with preserved ejection fraction. Eur J Heart Fail. 2011 Jan;13(1):18-28. doi: 10.1093/eurjhf/hfq121. Epub 2010 Aug 3. PMID 20685685
- [Background] Bhatia RS, Tu JV, Lee DS, Austin PC, Fang J, Haouzi A, Gong Y, Liu PP. Outcome of heart failure with preserved ejection fraction in a population-based study. N Engl J Med. 2006 Jul 20;355(3):260-9. doi: 10.1056/NEJMoa051530. PMID 16855266
- [Background] Owan TE, Hodge DO, Herges RM, Jacobsen SJ, Roger VL, Redfield MM. Trends in prevalence and outcome of heart failure with preserved ejection fraction. N Engl J Med. 2006 Jul 20;355(3):251-9. doi: 10.1056/NEJMoa052256. PMID 16855265
- [Background] McMurray JJ, Pfeffer MA. Heart failure. Lancet. 2005 May 28-Jun 3;365(9474):1877-89. doi: 10.1016/S0140-6736(05)66621-4. PMID 15924986
- [Background] NHFA CSANZ Heart Failure Guidelines Working Group; Atherton JJ, Sindone A, De Pasquale CG, Driscoll A, MacDonald PS, Hopper I, Kistler PM, Briffa T, Wong J, Abhayaratna W, Thomas L, Audehm R, Newton P, O'Loughlin J, Branagan M, Connell C. National Heart Foundation of Australia and Cardiac Society of Australia and New Zealand: Guidelines for the Prevention, Detection, and Management of Heart Failure in Australia 2018. Heart Lung Circ. 2018 Oct;27(10):1123-1208. doi: 10.1016/j.hlc.2018.06.1042. No abstract available. PMID 30077227
- [Background] Lewis GA, Schelbert EB, Williams SG, Cunnington C, Ahmed F, McDonagh TA, Miller CA. Biological Phenotypes of Heart Failure With Preserved Ejection Fraction. J Am Coll Cardiol. 2017 Oct 24;70(17):2186-2200. doi: 10.1016/j.jacc.2017.09.006. PMID 29050567
- [Background] Shah AM, Shah SJ, Anand IS, Sweitzer NK, O'Meara E, Heitner JF, Sopko G, Li G, Assmann SF, McKinlay SM, Pitt B, Pfeffer MA, Solomon SD; TOPCAT Investigators. Cardiac structure and function in heart failure with preserved ejection fraction: baseline findings from the echocardiographic study of the Treatment of Preserved Cardiac Function Heart Failure with an Aldosterone Antagonist trial. Circ Heart Fail. 2014 Jan;7(1):104-15. doi: 10.1161/CIRCHEARTFAILURE.113.000887. Epub 2013 Nov 18. PMID 24249049
- [Background] Persson H, Lonn E, Edner M, Baruch L, Lang CC, Morton JJ, Ostergren J, McKelvie RS; Investigators of the CHARM Echocardiographic Substudy-CHARMES. Diastolic dysfunction in heart failure with preserved systolic function: need for objective evidence:results from the CHARM Echocardiographic Substudy-CHARMES. J Am Coll Cardiol. 2007 Feb 13;49(6):687-94. doi: 10.1016/j.jacc.2006.08.062. Epub 2007 Jan 26. PMID 17291934
- [Background] Zile MR, Gottdiener JS, Hetzel SJ, McMurray JJ, Komajda M, McKelvie R, Baicu CF, Massie BM, Carson PE; I-PRESERVE Investigators. Prevalence and significance of alterations in cardiac structure and function in patients with heart failure and a preserved ejection fraction. Circulation. 2011 Dec 6;124(23):2491-501. doi: 10.1161/CIRCULATIONAHA.110.011031. Epub 2011 Nov 7. PMID 22064591
- [Background] Mohammed SF, Hussain S, Mirzoyev SA, Edwards WD, Maleszewski JJ, Redfield MM. Coronary microvascular rarefaction and myocardial fibrosis in heart failure with preserved ejection fraction. Circulation. 2015 Feb 10;131(6):550-9. doi: 10.1161/CIRCULATIONAHA.114.009625. Epub 2014 Dec 31. PMID 25552356
- [Background] Redfield MM. Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2016 Nov 10;375(19):1868-1877. doi: 10.1056/NEJMcp1511175. No abstract available. PMID 27959663
- [Background] Shah SJ, Lam CSP, Svedlund S, Saraste A, Hage C, Tan RS, Beussink-Nelson L, Ljung Faxen U, Fermer ML, Broberg MA, Gan LM, Lund LH. Prevalence and correlates of coronary microvascular dysfunction in heart failure with preserved ejection fraction: PROMIS-HFpEF. Eur Heart J. 2018 Oct 1;39(37):3439-3450. doi: 10.1093/eurheartj/ehy531. PMID 30165580
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982
- [Background] Arnold JR, Karamitsos TD, Bhamra-Ariza P, Francis JM, Searle N, Robson MD, Howells RK, Choudhury RP, Rimoldi OE, Camici PG, Banning AP, Neubauer S, Jerosch-Herold M, Selvanayagam JB. Myocardial oxygenation in coronary artery disease: insights from blood oxygen level-dependent magnetic resonance imaging at 3 tesla. J Am Coll Cardiol. 2012 May 29;59(22):1954-64. doi: 10.1016/j.jacc.2012.01.055. PMID 22624835
- [Background] Thulborn KR, Waterton JC, Matthews PM, Radda GK. Oxygenation dependence of the transverse relaxation time of water protons in whole blood at high field. Biochim Biophys Acta. 1982 Feb 2;714(2):265-70. doi: 10.1016/0304-4165(82)90333-6. PMID 6275909
- [Background] Karamitsos TD, Francis JM, Myerson S, Selvanayagam JB, Neubauer S. The role of cardiovascular magnetic resonance imaging in heart failure. J Am Coll Cardiol. 2009 Oct 6;54(15):1407-24. doi: 10.1016/j.jacc.2009.04.094. PMID 19796734
- [Background] Moon JC, Messroghli DR, Kellman P, Piechnik SK, Robson MD, Ugander M, Gatehouse PD, Arai AE, Friedrich MG, Neubauer S, Schulz-Menger J, Schelbert EB; Society for Cardiovascular Magnetic Resonance Imaging; Cardiovascular Magnetic Resonance Working Group of the European Society of Cardiology. Myocardial T1 mapping and extracellular volume quantification: a Society for Cardiovascular Magnetic Resonance (SCMR) and CMR Working Group of the European Society of Cardiology consensus statement. J Cardiovasc Magn Reson. 2013 Oct 14;15(1):92. doi: 10.1186/1532-429X-15-92. PMID 24124732
- [Background] Messroghli DR, Moon JC, Ferreira VM, Grosse-Wortmann L, He T, Kellman P, Mascherbauer J, Nezafat R, Salerno M, Schelbert EB, Taylor AJ, Thompson R, Ugander M, van Heeswijk RB, Friedrich MG. Clinical recommendations for cardiovascular magnetic resonance mapping of T1, T2, T2* and extracellular volume: A consensus statement by the Society for Cardiovascular Magnetic Resonance (SCMR) endorsed by the European Association for Cardiovascular Imaging (EACVI). J Cardiovasc Magn Reson. 2017 Oct 9;19(1):75. doi: 10.1186/s12968-017-0389-8. PMID 28992817
- [Background] Miller CA, Naish JH, Bishop P, Coutts G, Clark D, Zhao S, Ray SG, Yonan N, Williams SG, Flett AS, Moon JC, Greiser A, Parker GJ, Schmitt M. Comprehensive validation of cardiovascular magnetic resonance techniques for the assessment of myocardial extracellular volume. Circ Cardiovasc Imaging. 2013 May 1;6(3):373-83. doi: 10.1161/CIRCIMAGING.112.000192. Epub 2013 Apr 3. PMID 23553570
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. Circulation. 2017 Aug 8;136(6):e137-e161. doi: 10.1161/CIR.0000000000000509. Epub 2017 Apr 28. No abstract available. PMID 28455343
- [Background] D'Elia E, Vaduganathan M, Gori M, Gavazzi A, Butler J, Senni M. Role of biomarkers in cardiac structure phenotyping in heart failure with preserved ejection fraction: critical appraisal and practical use. Eur J Heart Fail. 2015 Dec;17(12):1231-9. doi: 10.1002/ejhf.430. Epub 2015 Oct 23. PMID 26493383
- [Background] Aronow WS, Ahn C, Kronzon I. Effect of propranolol versus no propranolol on total mortality plus nonfatal myocardial infarction in older patients with prior myocardial infarction, congestive heart failure, and left ventricular ejection fraction > or = 40% treated with diuretics plus angiotensin-converting enzyme inhibitors. Am J Cardiol. 1997 Jul 15;80(2):207-9. doi: 10.1016/s0002-9149(97)00320-2. PMID 9230162
- [Background] Setaro JF, Zaret BL, Schulman DS, Black HR, Soufer R. Usefulness of verapamil for congestive heart failure associated with abnormal left ventricular diastolic filling and normal left ventricular systolic performance. Am J Cardiol. 1990 Oct 15;66(12):981-6. doi: 10.1016/0002-9149(90)90937-v. PMID 2220622
- [Background] Cleland JG, Tendera M, Adamus J, Freemantle N, Polonski L, Taylor J; PEP-CHF Investigators. The perindopril in elderly people with chronic heart failure (PEP-CHF) study. Eur Heart J. 2006 Oct;27(19):2338-45. doi: 10.1093/eurheartj/ehl250. Epub 2006 Sep 8. PMID 16963472
- [Background] Yusuf S, Ostergren JB, Gerstein HC, Pfeffer MA, Swedberg K, Granger CB, Olofsson B, Probstfield J, McMurray JV; Candesartan in Heart Failure-Assessment of Reduction in Mortality and Morbidity Program Investigators. Effects of candesartan on the development of a new diagnosis of diabetes mellitus in patients with heart failure. Circulation. 2005 Jul 5;112(1):48-53. doi: 10.1161/CIRCULATIONAHA.104.528166. Epub 2005 Jun 27. PMID 15983242
- [Background] Massie BM, Carson PE, McMurray JJ, Komajda M, McKelvie R, Zile MR, Anderson S, Donovan M, Iverson E, Staiger C, Ptaszynska A; I-PRESERVE Investigators. Irbesartan in patients with heart failure and preserved ejection fraction. N Engl J Med. 2008 Dec 4;359(23):2456-67. doi: 10.1056/NEJMoa0805450. Epub 2008 Nov 11. PMID 19001508
- [Background] Shah RV, Desai AS, Givertz MM. The effect of renin-angiotensin system inhibitors on mortality and heart failure hospitalization in patients with heart failure and preserved ejection fraction: a systematic review and meta-analysis. J Card Fail. 2010 Mar;16(3):260-7. doi: 10.1016/j.cardfail.2009.11.007. Epub 2010 Jan 6. PMID 20206902
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Zile MR, O'Meara E, Claggett B, Prescott MF, Solomon SD, Swedberg K, Packer M, McMurray JJV, Shi V, Lefkowitz M, Rouleau J. Effects of Sacubitril/Valsartan on Biomarkers of Extracellular Matrix Regulation in Patients With HFrEF. J Am Coll Cardiol. 2019 Feb 26;73(7):795-806. doi: 10.1016/j.jacc.2018.11.042. PMID 30784673
- [Background] Solomon SD, Zile M, Pieske B, Voors A, Shah A, Kraigher-Krainer E, Shi V, Bransford T, Takeuchi M, Gong J, Lefkowitz M, Packer M, McMurray JJ; Prospective comparison of ARNI with ARB on Management Of heart failUre with preserved ejectioN fracTion (PARAMOUNT) Investigators. The angiotensin receptor neprilysin inhibitor LCZ696 in heart failure with preserved ejection fraction: a phase 2 double-blind randomised controlled trial. Lancet. 2012 Oct 20;380(9851):1387-95. doi: 10.1016/S0140-6736(12)61227-6. Epub 2012 Aug 26. PMID 22932717
- [Background] Diez J, Querejeta R, Lopez B, Gonzalez A, Larman M, Martinez Ubago JL. Losartan-dependent regression of myocardial fibrosis is associated with reduction of left ventricular chamber stiffness in hypertensive patients. Circulation. 2002 May 28;105(21):2512-7. doi: 10.1161/01.cir.0000017264.66561.3d. PMID 12034658
- [Background] Gori M, D'Elia E, Senni M. Sacubitril/valsartan therapeutic strategy in HFpEF: Clinical insights and perspectives. Int J Cardiol. 2019 Apr 15;281:158-165. doi: 10.1016/j.ijcard.2018.06.060. Epub 2018 Nov 9. PMID 30420146
- [Background] Sree Raman K, Nucifora G, Selvanayagam JB. Novel cardiovascular magnetic resonance oxygenation approaches in understanding pathophysiology of cardiac diseases. Clin Exp Pharmacol Physiol. 2018 May;45(5):475-480. doi: 10.1111/1440-1681.12916. Epub 2018 Feb 19. PMID 29350784
- [Background] Grover S, Lloyd R, Perry R, Lou PW, Haan E, Yeates L, Woodman R, Atherton JJ, Semsarian C, Selvanayagam JB. Assessment of myocardial oxygenation, strain, and diastology in MYBPC3-related hypertrophic cardiomyopathy: a cardiovascular magnetic resonance and echocardiography study. Eur Heart J Cardiovasc Imaging. 2019 Aug 1;20(8):932-938. doi: 10.1093/ehjci/jey220. PMID 30668650
- [Background] Chamsi-Pasha MA, Zhan Y, Debs D, Shah DJ. CMR in the Evaluation of Diastolic Dysfunction and Phenotyping of HFpEF: Current Role and Future Perspectives. JACC Cardiovasc Imaging. 2020 Jan;13(1 Pt 2):283-296. doi: 10.1016/j.jcmg.2019.02.031. Epub 2019 Jun 12. PMID 31202753
- [Background] Solomon SD, McMurray JJV, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, van Veldhuisen DJ, Zannad F, Zile MR, Desai AS, Claggett B, Jhund PS, Boytsov SA, Comin-Colet J, Cleland J, Dungen HD, Goncalvesova E, Katova T, Kerr Saraiva JF, Lelonek M, Merkely B, Senni M, Shah SJ, Zhou J, Rizkala AR, Gong J, Shi VC, Lefkowitz MP; PARAGON-HF Investigators and Committees. Angiotensin-Neprilysin Inhibition in Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2019 Oct 24;381(17):1609-1620. doi: 10.1056/NEJMoa1908655. Epub 2019 Sep 1. PMID 31475794
- [Background] Burke RM, Lighthouse JK, Mickelsen DM, Small EM. Sacubitril/Valsartan Decreases Cardiac Fibrosis in Left Ventricle Pressure Overload by Restoring PKG Signaling in Cardiac Fibroblasts. Circ Heart Fail. 2019 Apr;12(4):e005565. doi: 10.1161/CIRCHEARTFAILURE.118.005565. PMID 30998392